CLINICAL TRIAL: NCT00161239
Title: LAMPP Trial for Peripheral and Cutaneous T-Cell Lymphoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: toxicity
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Ortho Biotech, Inc. (Industry)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5192; CINJ#010410
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: T-Cell Lymphoma
Keywords: T-Cell Lymphomas
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — liposomal doxorubicin; Methotrexate; Asparaginase; Prednisone

INTERVENTIONS:
Drug: Doxil, Methotrexate, L-Asparaginase, Prednisone

SUMMARY:
Peripheral T cell lymphoma and advanced cutaneous T cell lymphomas are aggressive and refractory diseases that are generally treated with chemotherapy. Despite current treatment modalities, only a subset of patients will be cured by the treatment. In this study, four chemotherapeutic agents (L-asparaginase, Methotrexate, Doxil, and Prednisone) will be administered in a combination regimen for patients with relapsed or refractory Peripheral and/or advanced cutaneous T cell lymphoma. Each one of these individual drugs have been shown to have activity to lymphomas. The objective of the study is to determine if the combination of these chemotherapy agents results in higher response and cure rates in this patient population. This will be a single institutional study which will included 32 patients in the Peripheral T cell lymphoma group and 32 patients in the Cutaneous T cell lymphoma group.

DETAILED DESCRIPTION:
Peripheral T cell lymphoma and advanced cutaneous T cell lymphomas are aggressive and refractory diseases that are generally treated with chemotherapy. Despite current treatment modalities, only a subset of patients will be cured by the treatment. In this study, four chemotherapeutic agents (L-asparaginase, Methotrexate, Doxil, and Prednisone) will be administered in a combination regimen for patients with relapsed or refractory Peripheral and/or advanced cutaneous T cell lymphoma. Each one of these individual drugs have been shown to have activity to lymphomas. The objective of the study is to determine if the combination of these chemotherapy agents results in higher response and cure rates in this patient population. This will be a single institutional study which will included 32 patients in the Peripheral T cell lymphoma group and 32 patients in the Cutaneous T cell lymphoma group.

ELIGIBILITY:
Inclusion:

Patients must be at least 18 years of age. Histologically confirmed (including immunohistochemistry) diagnosis of T-Cell Lymphoma by skin biopsy or visceral/lymph node biopsy or bone marrow aspirate/biopsy Life expectancy of more than 3 months.

Exclusion:

Uncontrolled diabetes mellitus Active or serious infections uncontrolled with antibiotics Concurrent treatment, radiation or investigational treatment. 5.2.6 Significant underlying cardiac disease, including unstable angina, myocardial infarction less than 6 months before starting study, congestive failure of any cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2005-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of specific chemotherapy intervention

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, MD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Cancer Institute of New Jersey, New Brunswick, New Jersey, United States